CLINICAL TRIAL: NCT05327361
Title: Evaluation of the Depigmenting Effect of Liftactiv B3 Serum (Split Face) in Patients With Mild to Moderate Facial Post-acne PIHP for 3 Months
Brief Title: LiftActiv B3 in Post Inflammatory Hyperpigmentation (PIHP)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Enrollment timeline ended
Sponsor: University of Miami (Other)
Collaborators: Vichy Laboratoires (Industry)
Responsible Party: Principal Investigator, Leigh Nattkemper, Research Assistant Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20211099
Record Dates: First submitted 2022-03-14; First posted 2022-04-14 (Actual); Results first posted 2024-04-03 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-03

CONDITIONS: Acne; Post Inflammatory Hyperpigmentation
MeSH Terms: conditions — Acne Vulgaris; Hyperpigmentation | interventions — Sunscreening Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Group (Active Comparator): Participant will receive sunscreen in the morning and at the beginning of the afternoon for 3 months.
  Interventions: Other: Sunscreen
- Liftactiv B3 (Experimental): Participants will undergo a wash out phase of two weeks where they regularly apply a moisturizer (Hydreane Legere) in the morning and a sunscreen in the morning and at the beginning of the afternoon. On the 3rd week, participants will apply Liftactiv B3 serum daily in the morning before sunscreen and in the evening (two applications daily) on half face for 3 months.
  Interventions: Drug: Liftactiv B3

INTERVENTIONS:
Drug: Liftactiv B3 — Participants will apply a dime size amount of the serum to 1 side of the face.
  Arms: Liftactiv B3
Other: Sunscreen — Participants will apply a dime size amount of sunscreen to cover the other half of the face.
  Arms: Control Group

SUMMARY:
The purpose of this research study is to measure the depigmenting effect of a serum product called Liftactiv B3 in patients with mild to moderate facial PIHP (Post Inflammatory Hyper Pigmentation)

ELIGIBILITY:
Inclusion Criteria:

* Multiethnic subjects
* 18 to 50 YO
* Phototype III-VI
* All skin types
* 50% with sensitive skin (declarative)
* Symmetrical mild to moderate facial post-acne PIHP lesions with IGA scale
* Mild active acne (less than 10 retention and 5 inflammatory lesions)
* Agreeing not to change their lifestyle during the study period.
* Capable of reading the documents presented to them, of adhering to the study regulations and accepting the limitations.
* Available to follow the study
* Agreeing to participate and having signed the informed consent

Exclusion Criteria:

* Moderate to severe active acne
* Patients under topical or systemic retinoids
* Patients under systemic immunosuppressants
* Patients under active treatment of PIHP (including topicals or procedures) within the last 3 months
* Patients treated with facial procedures within the last 3 months
* Pregnancy
* Patient with a recent change in contraception (since less than 6 months)
* Known allergy to any component of tested product
* Not presenting with the conditions needed to comply with the protocol.
* Unable to give their informed consent
* Not available to follow the study in its entirety

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2022-03-22 (Actual); Primary Completion 2023-01-17 (Actual); Study Completion 2023-03-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Miami Hospital, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Every participant enrolled (total 13) received each arm of the study with treatment arm on one side of the face, and the control arm on the other side of the face (which equates to 26 "participants" total for the arms/groups).
Units Other Than Participants: Half face
Groups:
- All Study Participants: Participants will undergo a wash out phase of two weeks where they regularly apply a moisturizer (Hydreane Legere) in the morning and a sunscreen in the morning and at the beginning of the afternoon. On the 3rd week, participants will apply Liftactiv B3 serum daily in the morning before sunscreen and in the evening (two applications daily) on half face for 3 months.
  Liftactiv B3: Participants will apply a dime size amount of the serum to 1 side of the face.
  Sunscreen: Participants will apply a dime size amount of sunscreen to cover the other half of the face.
  Participant will receive sunscreen in the morning and at the beginning of the afternoon for 3 months.
Period: Overall Study
Arm/Group | All Study Participants
Started | 13; 26 Half face
Liftactiv B3 | 13; 26 Half face
Control Group | 13; 26 Half face
Completed | 9; 18 Half face
Not Completed | 4; 8 Half face
Not completed — Lost to Follow-up | 4

BASELINE CHARACTERISTICS:
Groups:
- Liftactiv B3 and Control Group: Participants will undergo a wash out phase of two weeks where they regularly apply a moisturizer (Hydreane Legere) in the morning and a sunscreen in the morning and at the beginning of the afternoon. On the 3rd week, participants will apply Liftactiv B3 serum daily in the morning before sunscreen and in the evening (two applications daily) on half face for 3 months.
  Liftactiv B3: Participants will apply a dime size amount of the serum to 1 side of the face.
  Sunscreen: Participants will apply a dime size amount of sunscreen to cover the other half of the face.
  Participant will receive sunscreen in the morning and at the beginning of the afternoon for 3 months.will apply a dime size amount of sunscreen to cover the other half of the face.
Arm/Group | Liftactiv B3 and Control Group
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 5
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Post Inflammatory Hyperpigmentation (PIHP) Change
Description: Post Inflammatory Hyperpigmentation (PIHP) will be evaluated using the post acne hyperpigmentation scale.
  The total score can range from 6-22 points. Subscales will measure lesion size, lesion intensity, and number of lesions. Subscales are added together to form the total score. Higher values indicate worse hyperpigmentation.
Time Frame: Baseline, 1 month, 2 months and 3 months
Population: Only 9 participants completed the the follow up (1 month, 2 month, and 3 month) visit assessments.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Group | Liftactiv B3
Number analyzed (Participants) | 9 | 9
score on a scale
  Baseline | 8.25 (2.38) | 8.25 (2.37)
  1 month | 6.56 (1.13) | 6.56 (1.13)
  2 months | 6.44 (1.33) | 6.44 (1.33)
  3 months | 6 (0) | 6 (0)

2. Secondary Outcome: Change in the Investigators Global Assessment (IGA) Scale
Description: Pigmentation will also be evaluated clinically using the Physician global assessment IGA defined as clear is 0, almost clear is 1, mild is 2, moderate is 3, severe is 4, and every severe is 5 within the treatment area.
Time Frame: Baseline, 1 month, 2 months and 3 months
Population: Only 12 participants completed the follow up (1 month, 2 month, and 3 month) visit assessments.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control Group | Liftactiv B3
Number analyzed (Participants) | 9 | 9
units on a scale
  Baseline | 2.08 (0.79) | 1.92 (0.79)
  1 month | 1.33 (0.5) | 1.22 (0.44)
  2 months | 1.33 (0.87) | 1.33 (0.87)
  3 months | 1.33 (0.87) | 1.44 (0.88)

3. Secondary Outcome: Change in Skin Condition Evaluation Scores
Description: Clinical evaluation of skin condition on subject's face which includes deep wrinkles, fine lines, skin tone, skin texture, radiance and skin elasticity will be evaluated using a 10 point Likert Scale. Each of these conditions will use the same Likert Scale from 0 to 9 with the higher score indicating more severe/worse symptoms.
Time Frame: Baseline, 1 month, 2 months and 3 months
Population: Only 9 participants completed the the follow up (to 3 month) visit assessments. Oversight of translation from protocol to CRF caused this data to not be collected at 1month and 2 month time points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control Group | Liftactiv B3
Number analyzed (Participants) | 9 | 9
units on a scale
  3 months | 4.44 (1.57) | 2.67 (1.33)
  2 months: number analyzed (Participants) | 0 | 0
  1 months: number analyzed (Participants) | 0 | 0
  Baseline | 5.33 (1.33) | 5.33 (1.33)

4. Secondary Outcome: Change in Global Efficacy Assessment
Description: Global efficacy of the treatment evaluated at each visit by the patient.
  The measure of the global efficacy will be realized according to the Global efficacy scale which ranges from nil to excellent which will be measured from 0 (equals nil) to 4 (equals excellent).
Time Frame: 1 month, 2 months, and 3 months
Population: as for outcome 3
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | All Study Participants
Number analyzed (Participants) | 9
score on a scale
  3 months | 2.56 (0.68)
  2 months: number analyzed (Participants) | 0
  1 month: number analyzed (Participants) | 0

5. Secondary Outcome: Change in Global Tolerance Score
Description: Clinical tolerance global score will be assessed, on the treated area, at each visit using first a 4-point skin reaction scale which ranges from 0 which indicates no evidence of local intolerance and 4 indicates very severe signs or symptoms of intolerance.
Time Frame: 1 month, 2 months, and 3 months
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Study Participants
Number analyzed (Participants) | 9
score on a scale
  3 months | 0.11 (0.31)
  2 months: number analyzed (Participants) | 0
  1 month: number analyzed (Participants) | 0

6. Secondary Outcome: Change in Cosmeticity Questionnaire and Acceptability
Description: Subjects will be questioned about their perceived effects of the investigational product on their skin.
  The cosmeticity questionnaire is a 5 point scale (1-fully disagree; 2-disagree partly; 3-no opinion; 4-agree partly; 5-fully agree).
Time Frame: 1 month, 2 months, and 3 months
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Study Participants
Number analyzed (Participants) | 9
score on a scale
  3 months | 4.39 (0.5)
  2 months: number analyzed (Participants) | 0
  1 month: number analyzed (Participants) | 0

7. Secondary Outcome: Exposome Questionnaire
Description: Subjects will be questioned about environmental influences. Count of participants completing questionnaire.
Time Frame: Baseline and 3 months
Population: Exposome questionnaire only consists of descriptive questions (used for data collection only), so reported here as number of participants that completed questionnaire.
Measure: Count of Participants; unit: Participants
Arm/Group | All Study Participants
Number analyzed (Participants) | 9
Participants
  3 months | 9
  Baseline | 9

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Control Group | Liftactiv B3
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 0/13 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-14): https://cdn.clinicaltrials.gov/large-docs/61/NCT05327361/Prot_SAP_000.pdf